CLINICAL TRIAL: NCT03391856
Title: A Prospective Randomized Controlled Study for Intervention of Prolonged Isolated Thrombocytopenia After Allogeneic Hematopoietic Stem Cell Transplantation: N-acetyl-L-cysteine (NAC) Versus Supportive Therapy
Brief Title: Prolonged Isolated Thrombocytopenia After Allo-SCT : N-acetyl-L-cysteine (NAC) Versus Supportive Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: protocol changed
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Head of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017PHB220
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Thrombocytopenia; Stem Cell Transplant Complications
MeSH Terms: conditions — Thrombocytopenia | interventions — Acetylcysteine; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): NAC 400mg p.o tid from day 60 to day 90 post transplant
  Interventions: Drug: N-acetyl-L-cysteine (NAC)
- controlled arm (Other): Supportive therapy including platelet infusion:prophylactic platelet transfusion was given when platelet count <20000/ul
  Interventions: Other: supportive therapy

INTERVENTIONS:
Drug: N-acetyl-L-cysteine (NAC) — NAC treatment for PT: 400mg p.o tid from day 60 to 90 post transplant
  Arms: intervention arm
Other: supportive therapy — prophylactic platelet transfusion was given when platelet count <20000/ul
  Arms: controlled arm

SUMMARY:
Isolated prolonged thrombocytopenia (PT) is a common complication after allogeneic stem cell transplantation with significant poor prognosis. No standard treatment is available. The current study assigned PT randomly to 2 arms: intervention arm with N-acetyl-L-cysteine (NAC) and control arm with supportive therapy.This is a prospective randomized controlled study.

DETAILED DESCRIPTION:
1. patients diagnosed with PT at day 60 post transplant will be randomized assigned to intervention arm (NAC) or controlled arm (supportive therapy: prophylactic platelet transfusion was given when platelet count <20000/ul.)
2. Response will be evaluated at day 90. Response was defined as platelet recovery to >= 20000/ul for 7 consecutive days without transfusion support during the enrollment period. All the other patients not achieved above criteria was defined as no response.
3. For those without response in both arms, patients will received NAC plus recombinant human thrombopoietin (rhTPO) for an additional 30 days. rhTPO was given at 300IU/kg/d for 28 consecutive days or platelet > 50000/ul independent of platelet transfusion.

ELIGIBILITY:
Inclusion Criteria:

* age>= 14 years
* diagnosed as PT (defined as platelet count in peripheral blood never achieve 20000/miro-liter for 7 consecutive days without transfusion at day 60 post transplantation)
* serum creatine level < ULN (upper limit of normal), serum ALT/AST /TBil<=2 ULN
* without active CMV/EBV/ADV reactivation, active GVHD, without relapse or minimal residual disease at enrollment

Exclusion Criteria:

* history of asthma
* allergy to NAC
* refuse to participate

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
response rate | 30 days after the start of enrollement
  rate of response after 30 days of treatment

SECONDARY OUTCOMES:
overall survival | the day of last follow-up
  survival proportion at the last followup after transplantation
non-relapse mortality | the day of last follow-up
  non-relapse mortality at the last followup after transplantation
grade 2-4 acute graft versus host disease | day 100 after transplant
  grade 2-4 aGVHD at day 100 after transplant
chronic graft versus host disease | the day of last follow-up
  chronic graft versus host disease at the day of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peiking University
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No